CLINICAL TRIAL: NCT04961996
Title: A Phase III, Randomized, Open-Label, Multicenter Study Evaluating the Efficacy and Safety of Adjuvant Giredestrant Compared With Physician's Choice of Adjuvant Endocrine Monotherapy in Patients With Estrogen Receptor-Positive, HER2-Negative Early Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Adjuvant Giredestrant Compared With Physician's Choice of Adjuvant Endocrine Monotherapy in Participants With Estrogen Receptor-Positive, HER2-Negative Early Breast Cancer (lidERA Breast Cancer)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42784; 2021-000129-28 (EudraCT Number); 2023-507172-44-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Gonadotropin-Releasing Hormone; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Giredestrant (Experimental)
  Interventions: Drug: Giredestrant; Drug: LHRH Agonist
- Arm B: Endocrine Therapy of Physician's Choice (Active Comparator)
  Interventions: Drug: Endocrine Therapy of Physician's Choice; Drug: LHRH Agonist
- Substudy: Giredestrant + Abemaciclib, Then Giredestrant (Experimental): In this substudy, participants will receive giredestrant in combination with abemaciclib for up to 2 years. Participants will continue with giredestrant monotherapy for an additional 3 years in order to complete a total of 5 years on study treatment.
  Interventions: Drug: Giredestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Giredestrant — Giredestrant 30 milligrams (mg) will be administered orally once a day (QD) on Days 1-28 of each 28-day cycle for 5 years or until disease recurrence or unacceptable toxicity (whichever occurs first).
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Arm A: Giredestrant; Substudy: Giredestrant + Abemaciclib, Then Giredestrant
Drug: Endocrine Therapy of Physician's Choice — The endocrine therapy of physician's choice (TPC) is limited to tamoxifen or one of the specified third generation aromatase inhibitors: letrozole, anastrozole, or exemestane. Participants will receive TPC daily on Days 1-28 of each 28-day cycle for 5 years or until disease recurrence or unacceptable toxicity (whichever occurs first). Continuing TPC after 5 years is at the discretion of the investigator and per local standard of care. Dose administration of TPC should be performed in accordance with the local prescribing information for the respective product.
  Arms: Arm B: Endocrine Therapy of Physician's Choice
Drug: LHRH Agonist — A luteinizing hormone-releasing hormone (LHRH) agonist will be administered to male participants and premenopausal/perimenopausal participants according to local prescribing information. The investigator may determine and supply the appropriate LHRH agonist locally approved for use in breast cancer.
  Arms: Arm A: Giredestrant; Arm B: Endocrine Therapy of Physician's Choice
Drug: Abemaciclib — Abemaciclib 150 mg will be administered orally (PO) twice a day (BID) on Days 1-28 during each 28-day cycle for 2 years or until disease recurrence or unacceptable toxicity (whichever occurs first).
  Arms: Substudy: Giredestrant + Abemaciclib, Then Giredestrant

SUMMARY:
This is a Phase III, global, randomized, open-label, multicenter, study evaluating the efficacy and safety of adjuvant giredestrant compared with endocrine therapy of physician's choice in participants with medium- and high-risk Stage I-III histologically confirmed estrogen receptor (ER)-positive and human epidermal growth factor receptor 2 (HER2)-negative early breast cancer.

In addition, an open-label exploratory substudy will explore the safety and efficacy of giredestrant in combination with abemaciclib in a subset of the primary study population.

ELIGIBILITY:
Primary Study Inclusion Criteria:

* Documented estrogen receptor (ER)-positive and HER2-negative breast tumor, as assessed locally on a primary disease specimen
* Participants who have multicentric (the presence of two of more tumor foci within different quadrants of the same breast) and/or multifocal (the presence of two or more tumor foci within a single quadrant of the breast) breast cancer are also eligible if all examined tumors meet pathologic criteria for ER positivity and HER2 negativity
* Participants must have undergone definitive surgery of their primary breast tumor(s) and axillary lymph nodes (axillary lymph node dissection [ALND] and/or sentinel lymph node biopsy [SLNB])
* Participants who received or will be receiving adjuvant chemotherapy must have completed adjuvant chemotherapy prior to randomization. Participants may also have received neoadjuvant chemotherapy. A washout period of at least 21 days is required between last adjuvant chemotherapy dose and randomization.
* Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE v5.0 Grade 1 or better (except alopecia, Grade ≤2 peripheral neuropathy, arthralgia or other toxicities not considered a safety risk for the participant per the investigator's judgment)
* Participants have received (neo)adjuvant chemotherapy and/or had surgery and had no prior endocrine therapy are eligible, provided that they are enrolled within 12 months following definitive breast cancer surgery
* Participants who have confirmed availability of an untreated primary breast tumor tissue specimen suitable for biomarker testing (i.e., representative archived formalin-fixed, paraffin-embedded [FFPE] tissue block [preferred] or 15-20 slides containing unstained, freshly cut, serial sections), with associated de-identified pathology report is required. Although 15-20 slides are preferred, if only 10-14 slides are available, the individual may still be eligible for the study.
* Participants with node-positive and node-negative disease are eligible provided they meet additional risk criteria as defined in the protocol
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2
* Able and willing to swallow, retain, and absorb oral medication
* Adequate organ function

Substudy Inclusion Criteria:

To be eligible for substudy participation, in addition to meeting the inclusion criteria in the primary protocol, participants must also meet the following modified criteria:

- Patients who received adjuvant radiotherapy must have completed radiotherapy prior to enrollment, and patients must have recovered (to Grade ≤1) from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and enrollment.

Primary Study Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 10 days after the final dose of giredestrant, or within the time period specified per local prescribing guidelines after the final dose of the endocrine therapy of physician's choice
* Received treatment with investigational therapy within 28 days prior to initiation of study treatment or is currently enrolled in any other type of medical research judged by the sponsor not to be scientifically or medically compatible with this study
* Receiving or planning to receive a CDK4/6 inhibitor as (neo)adjuvant therapy. A short course of up to 12 weeks of neoadjuvant or adjuvant treatment with CDK4/6 inhibitor therapy prior to randomization is allowed.
* Active cardiac disease or history of cardiac dysfunction
* Diagnosed with Stage IV breast cancer
* A history of any prior (ipsilateral and/or contralateral) invasive breast cancer or ductal carcinoma in situ (DCIS). Participants with a history of contralateral DCIS treated by only local regional therapy at any time may be eligible.
* A history of any other malignancy within 3 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, or Stage I uterine cancer
* Any prior endocrine treatment with selective ER modulators (e.g., tamoxifen), degraders, or aromatase inhibitors. A short course of neoadjuvant or adjuvant endocrine therapy (up to 12 weeks) is allowed.
* Clinically significant liver disease consistent with Child-Pugh Class B or C, including active hepatitis (e.g., hepatitis B virus [HBV] or hepatitis C virus [HCV]), current alcohol abuse, cirrhosis, or positive test for viral hepatitis
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients
* Pre- and perimenopausal participants or male participants who have a known hypersensitivity to LHRH agonists
* A documented history of hemorrhagic diathesis, coagulopathy, or thromboembolism
* Renal dysfunction that requires dialysis
* A major surgical procedure unrelated to breast cancer within 28 days prior to randomization
* A serious infection requiring oral or IV antibiotics within 14 days prior to screening or other clinically significant infection (e.g., COVID-19) within 14 days prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes an individual's safe participation in and completion of the study
* Unable or unwilling to comply with the requirements of the protocol in the opinion of the investigator

Substudy Exclusion Criteria:

Potential participants are excluded from the substudy if any criteria from t\he primary study or the following criteria apply:

* Prior participation in the GO42784 primary study
* Received a CDK4/6i as (neo)adjuvant therapy prior to enrollment
* Treatment with moderate CYP3A inducers, strong CYP3A inducers or strong CYP3A inhibitors within 14 days or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS), Excluding Second Primary Non-Breast Cancers | From randomization to first occurrence of an IDFS event (up to 10 years)

SECONDARY OUTCOMES:
Overall Survival | From randomization to death from any cause (up to 10 years)
Invasive Disease-Free Survival (IDFS), Including Second Primary Non-Breast Cancers | From randomization to first occurrence of an IDFS event (up to 10 years)
Disease-Free Survival (DFS) | From randomization to first occurrence of a DFS event (up to 10 years)
Distant Recurrence-Free Interval (DRFI) | From randomization to first occurrence of a DFRI event (up to 10 years)
Locoregional Recurrence-Free Interval (LRRFI) | From randomization to first occurrence of a LRRFI event (up to 10 years)
Mean Physical Functioning Scale Score at Specified Timepoints, Assessed Using the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Change from Baseline in the Mean Physical Functioning Scale Score at Specified Timepoints, Assessed Using the EORTC QLQ-C30 | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Mean Role Functioning Scale Score at Specified Timepoints, Assessed Using the EORTC QLQ-C30 | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Change from Baseline in the Mean Role Functioning Scale Score at Specified Timepoints, Assessed Using the EORTC QLQ-C30 | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Mean Global Health Status/Quality of Life (QoL) Scale Score at Specified Timepoints, Assessed Using the EORTC QLQ-C30 | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Change from Baseline in the Mean Global Health Status/Quality of Life (QoL) Scale Score at Specified Timepoints, Assessed Using the EORTC QLQ-C30 | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Change from Baseline in the EQ 5D-5L Index-Based Score at Specified Timepoints | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Change from Baseline in the EQ 5D-5L Visual Analogue Scale (VAS) Score at Specified Timepoints | Baseline (Cycle 1) and Cycles 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, and 60 (1 cycle is 28 days) of treatment, once every 6 months during the first 2 years of post-treatment follow-up and annually for 3 years thereafter (up to 10 years)
Incidence and Severity of Adverse Events, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | From start of treatment until 28 days after the final dose of study treatment (up to 5 years)
Plasma Concentrations of Giredestrant at Specified Timepoints | Predose and 3-4 hours postdose on Day 1 of Cycles 1 and 2, and predose on Day 1 of Cycles 3 and 6 (1 cycle is 28 days)
Substudy: Incidence of Grade ≥3 Adverse Events with Giredestrant in Combination with Abemaciclib | From first dose of study treatment until 28 days after the last dose of treatment with the combination of giredestrant and abemaciclib or until the end of Year 2, whichever occurs first (up to 2 years)
Substudy: Incidence and Severity of Adverse Events with Giredestrant in Combination with Abemaciclib, with Severity Determined According to NCI-CTCAE v5.0 | From first dose of study treatment until 28 days after the last dose of treatment with the combination of giredestrant and abemaciclib or until the end of Year 2, whichever occurs first (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (627):
- United States (86):
  - Southern Cancer Center, Daphne, Alabama
  - CBCC Global Research Inc., at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Arrowhead Regional Medical Center, Colton, California
  - Cancer and Blood Specialty Clinic, Fountain Valley, California
  - St Joseph Heritage Healthcare, Fullerton, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Keck Medicine of USC ? Newport Beach, Newport Beach, California
  - The Center for Cancer Prevention and Treatment at St.Joseph Hospital of Orange, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Kaiser Permanente - San Diego, San Diego, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Sansum Clinic, Santa Barbara, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Torrance Memorial Physician Network/Cancer Care, Torrance, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Rocky Mountain Cancer Centers (Longmont) - USOR, Longmont, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System - Memorial Regional Hospital, Hollywood, Florida
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Miami Cancer Institute-Plantation, Plantation, Florida
  - Memorial Health University Cancer Center, Savannah, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Elmhurst Cancer Center, Elmhurst, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - Duly Health and Care, Tinley Park, Illinois
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute - MDC, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - UPMC Western Maryland - Schwab Family Cancer Center, Cumberland, Maryland
  - University of Maryland, Towson, Maryland
  - Lahey Clinic Med Ctr, Burlington, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - University of Missouri-Columbia, Columbia, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Cancer Cen, New York, New York
  - Stony Brook Univ Cancer Ctr, Stony Brook, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Kaiser Permanente-Northwest Region, Portland, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Penn State Univ. Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - Texas Oncology, P.A. - El Paso, El Paso, Texas
  - Texas Oncology (Flower Mound) - USOR, Flower Mound, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Texas Oncology (McAllen) - USOR, McAllen, Texas
  - Texas Oncology McKinney, McKinney, Texas
  - Texas Oncology (Tyler) - USOR, Tyler, Texas
  - Texas Oncology (Waco) - USOR, Waco, Texas
  - Centra Alan B. Pearson Regional Cancer Center, Lynchburg, Virginia
  - Bon Secours Mercy Health, Midlothian, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc.,-Blacksburg, Roanoke, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (23):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Fundacion Intectus, Bariloche, Río Negro Province
  - Hospital Italiano Regional del Sur, Bahía Blanca
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Metabólicas (IDIM), Buenos Aires
  - Centro Oncologico Korben, Caba
  - Fundacion Medica de Rio Negro Y Nuequen, Cipolletti
  - Consultorios Médicos Dr. Doreski, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende Servicio Nefrología, Córdoba
  - Centro Medico Privado CEMAIC, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Hospital Privado de La Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - Instituto de Especialidades de la Salud Rosario - Clínica del Tórax, Rosario
  - Sanatorio Parque de Rosario, Rosario
  - Instituto de Oncologia de Rosario, Rosario
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
  - Centro Medico San Roque, San Miguel de Tucumán
  - Organizacion Medica de Investigacion, San Nicolás
  - Fundación Ars Medica, San Salvador de Jujuy
  - Centro de Investigación Clínica ? Clínica Viedma, Viedma
- Australia (21):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Northmead, New South Wales
  - Mater Hospital, Wollstonecraft, New South Wales
  - Mater Cancer Care Centre, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Andrews Medical Centre, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - ICON Cancer Care Hobart, Hobart, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Northern Hospital, Epping, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - South West Healthcare, Warrnambool, Victoria
  - Ballarat Oncology & Haematology, Wendouree, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (9):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH, Linz
  - LKH Rankweil, Interne E, Rankweil
  - Universitätsklinikum Salzburg, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - A.ö. Krankenhaus der Barmherzigen Brüder, Sankt Veit im Pongau
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
  - Medizinische Universitat Wien Medical University of Vienna, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (10):
  - Institute Jules Bordet, Belgium
  - Grand Hopital de Charleroi asbl, Charleroi
  - UZ Leuven, Leuven
  - CH de l'Ardenne (Libramont), Libramont
  - Centre Hospitalier Chrétien MontLégia, Liège
  - CHR de la Citadelle, Pharmacie, Liège
  - Chu Sart Tilman, Liège
  - Clinique Sainte-Elisabeth, Namur
  - Cliniques Universitaires UCL de Mont-Godinne, Namur
  - GZA Ziekenhuizen Antwerpen campus Sint-Augustinus, Wilrijk
- Bosnia and Herzegovina (3):
  - Clinical Center Banja Luka, Banja Luka
  - Clinical Hospital Mostar, Mostar
  - University Clinical Center Tuzla, Tuzla
- Brazil (26):
  - Centro Odonito Medico Linus Pauling - Clinica de O, Salvador, Estado de Bahia
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - Centro de Oncologia da Bahia, Salvador/BA, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Cenantron - Centro Avancado de Tratamento Oncologico, Belo Horizonte, Minas Gerais
  - Oncoclinicas do Brasil Servicos Medicos As, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Pôrto Alegre, Pará
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Universidade de Caxias do Sul - Rio Grande do Sul, Caixas Do Sul, Rio Grande do Sul
  - ONCOSITE Centro de Pesquisa Clínica Em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Vicente de Paulo X, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - *X*Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto de Oncologia Clínica de Piracicaba, Piracicaba, São Paulo
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
  - Clinica de Pesquisas e Centro de Estudos Oncologia Ginecologica e Mamaria Ltda, São Paulo
  - Onco Star Sp Oncologia Ltda, São Paulo
- Bulgaria (2):
  - Complex Oncology Center Burgas, Burgas
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
- Canada (15):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Centre Integre Universitaire de Sante et de Services Sociaux du Saguenay Lac Saint Jean, Chicoutimi, Quebec
  - Hopital Charles Le Moyne, Greenfield Park, Quebec
  - CIUSSS-de-l?Est-de-l?Île-de-Montréal, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - St-Jérome Medical Research, Inc., Saint-Jérôme, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - CHU de Quebec-Universite Laval, Québec
- Chile (12):
  - Fundacion Arturo Lopez Perez (FALP) - Providencia - Jose Manuel Infante 805, Providencia, Región-MetropolitanadeSantiago
  - IC La Serena Research SpA, La Serena
  - Patagonia Research, Port Montt
  - Centro de Estudios Clínicos SAGA SpA, Providencia
  - Servicios Médicos URUMED SpA, Rancagua
  - Oncovida - Santiago, Santiago
  - Centro de Estudios Clinicos E Investigaciones Medicas, Santiago
  - Icegclinic, Santiago
  - Medwal, Santiago
  - James Lind Centro de Investigación Del Cáncer, Temuco
  - Oncocentro Apys, Viña del Mar
  - Centro de Investigaciones Clinicas Viña del Mar, Viña del Mar
- China (34):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University People's Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Guangdong Provincial Maternity and Child Care Cent, Guangzhou
  - Sun yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Cancer Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Linyishi Cancer Hospital, Linyi
  - The Third Hospital of Nanchang, Nanchang
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Wenzhou Medical College - The First Affiliated Hospital GCP, Wenzhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Air Force Military Medical University Xijing Hospital, Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
- Colombia (3):
  - Oncomedica S.A., Montería, Departamento de Córdoba
  - Hemato Oncólogos S.A, Cali
  - FOSCAL, Floridablanca
- Costa Rica (4):
  - Consultorio Oncologico-Hospital Metropolitano Linc, Moravia
  - Metropolitano Research Institute Lindora, San José
  - Centro de Cáncer y Hematología, San José
  - Instituto de Investigación en Ciencias Médicas S.A., San José
- Croatia (6):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - University Hospital of Split, Split
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Sestre Milosrdnice, Zagreb
  - Klinicki bolnicki centar Zagreb, Zagreb
- Czechia (4):
  - Fakultni nemocnice Olomouc, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova Nemocnice, Prague
- Egypt (7):
  - Mansoura University Hospital, Al Mansurah
  - Alexandria Uni, Alexandria
  - Medical Technology Center for Research and Services, Alexandria
  - Kasr Al Ainy School of Medicine-Cairo University, Cairo
  - Ain Shams University Hospital, Cairo
  - Gustave Roussy International Egypt Hospital, Fostat
  - Sohag Oncology Center, Markaz Sohag
- Finland (3):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun Yliopistollinen Keskussairaala, Turku
- France (23):
  - Centre Francois Baclesse, Caen, Calvados
  - Clinique Clémentville, Montpellier, Hérault
  - Sas Clinique De L Europe - Amiens, Amiens
  - Hopital d'Argenteuil, Argenteuil
  - Centre Hospitalier Regional Universitaire de Brest - Hopital de la Cavale Blanche, Brest
  - Institut Daniel Hollard, Grenoble
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre de cancérologie de la Sarthe - Aile B, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Privé Clairval, Marseille
  - Clinique Catherine de Sienne, Nantes
  - Hopital Universitaire Pitie Salpetriere, Paris
  - Hopital Tenon, Paris
  - Institut Curie, Paris
  - Hopital Saint Louis, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital privé des Côtes Armor, Plérin
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes
  - Centre Henri Becquerel, Rouen
  - Curie Saint Cloud, Saint-Cloud
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Georgia (7):
  - High Technology Hospital MedCenter Ltd, Batumi
  - Acad. F. Todua Medical Center, Tbilisi
  - Ltd Israel-Georgia Medical Research Clinic Helsicore, Tbilisi
  - LTD Health House, Tbilisi
  - Institute of Clinical Oncology LTD, Tbilisi
  - LTD TIM, Tbilisi Institute of Medicine, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (18):
  - Hämatologisch/onkologische Gemeinschaftspraxis, Augsburg
  - Ambulantes Tumorzentrum Spandau, Berlin
  - Lübecker Onkologische Schwerpunktpraxis, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Erlangen, Erlangen
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Franziskus-Hospital Harderberg, Georgsmarienhütte
  - SRH Wald-Klinikum Gera, Gera
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Gynäkologisch Onkologische Praxis Hannover, Hanover
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Facharztpraxis für Gynäkologie und Geburtshilfe PD Dr. med. Christian Kurbacher, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Praxis fuer gynaekologische onkologie Prof. Dr. me, Mönchengladbach
  - Hämatologie und Onkologie Ravensburg / Wangen, Ravensburg
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt
  - Praxis fur Haematologie und Internistische Onkologie, Velbert
- Greece (20):
  - European Interbalkan Medical Center, Pylaia, Thessaloniki
  - Henry Dunant Hospital, Athens
  - University of Athens, Hematological Clinic,, Athens
  - Aretaieio Hospital of Athens, Athens
  - Sotiria Chest Hospital of Athens, Athens
  - General Oncology Hospital Kifissias "Oi Agioi Anargyroi", Athens
  - Attikon University General Hospital, Chaïdári
  - Metropolitan General Hospital, Cholargós
  - Metropolitan Hospital First Oncology Clinic, Faliro
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - IASO Obstetrics Gynecology Clinic, Marousi
  - Medical Center of Athens, Marousi
  - Olympion Clinic, Pátrai
  - University General Hospital of Patras, Pátrai
  - Bioclinic Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - St. Luke's Hospital, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Guatemala (5):
  - Celan S.A., Guatemala City
  - INTEGRA Cancer Institute, Guatemala City
  - Oncomedica, Guatemala City
  - Grupo Medico Angeles, Guatemala City
  - Clínica Médica Especializada en Hematología, Guatemala City
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (7):
  - Semmelweis Egyetem, Budapest
  - Tolna Megyei Balassa János Kórház, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szent Borbala Korhaz, Tatabánya
  - Zala Megyei Szent Rafael Korhaz, Zalaegersteg
- India (20):
  - HCG City Cancer Centre, Vijayawada, Andhra Pradesh
  - State Cancer Institute, Indira Gandhi Institute of Medical Sciences (IGIMS), Patna, Bihar
  - Nirmal Hospital, Surat, Gujarat
  - Kiran Hospital Multi Super Speciality Hospital and Research Center, Surat, Gujarat
  - Himalaya Cancer Hospital & Research Institute, Vadodara, Gujarat
  - Kailash Cancer Hospital and Research Center, Vadodara, Gujarat
  - KLES Dr Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Sujan Surgical Cancer Hospital And Amravati Cancer Foundation, Amravati, Maharashtra
  - Kolhapur Cancer Centre, Kolhāpur, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Government Medical College, Nagpur, Maharashtra
  - Shalinitai Meghe Medical College and Hospital, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Chopda Medicare & Research Centre pvt. Ltd, Nashik, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Specialty Hospital Hadapsar, Pune, Maharashtra
  - Lokmanya Holistic Cancer Care and Research Center (LMRC), Pune, Maharashtra
  - Erode Cancer Centre, Erode, Tamil Nadu
  - Christian Medical College-Ranipet Campus, Ratnagiri Kilminnal, Tamil Nadu
- Ireland (7):
  - Cork University Hospital, Cork
  - Bon Secours Hospital, Cork
  - St Vincents University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
  - Mid- Western Regional Hospital Limerick, Limerick
  - Waterford Regional Hospital, Waterford
- Israel (3):
  - Soroka University Medical Centre, Beersheba
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Roma, Emilia-Romagna
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Ospedale San Giuseppe, Empoli, Tuscany
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Usl Toscana nord ovest - Ospedali Riuniti di Livorno, Livorno, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
- Japan (12):
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima University Hospital, Hiroshima
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - Saitama Cancer Center, Kitaadachi-gun
  - Kumamoto University Hospital, Kumamoto-Shi Chuo-Ku
  - Nahanishi Clinic, Naha
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - St. Luke's International Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
- Kenya (2):
  - International Cancer Institute (ICI), Eldoret
  - The Aga Khan University-Kenya., Nairobi
- Pauls Stradins Clinical University Hospital, R?ga, Latvia
- Malaysia (7):
  - Hospital Kuala Lumpur, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - National Cancer Institute IKN, Putrajaya, Federal Territory of Putrajaya
  - Pantai Hospital Sungai Petani, Sungai Petani, Kedah
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Sarawak General Hospital, Buzia?, Sarawak
  - Beacon International Specialist Centre, Petaling Jaya, Selangor, Selangor
- Mexico (17):
  - Centro de Investigación en Artritis y Osteoporosis - PPDS, Mexicali, Estado de Baja California
  - Dr. José Luis González Trujillo, León, Guanajuato
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Clínica Integral Internacional de Oncología S de RL de CV, Puebla City, Mexico CITY (federal District)
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Investigación Médica de Alta Especialidad, Querétaro City, Querétaro
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Merida | Investigacion Clinica, Mérida, Yucatán
  - Centro de Investigacion Medica Aguascalientes, Aguascalientes
  - Centro Oncologico Alianza XXI, México
  - Oaxaca Site Management Organization, Oaxaca City
  - Oncologica de Puebla S.A de C.V, Puebla City
  - Oncológico Potosino, San Luis Potosí City
  - Centro Hemato-Oncologico Privado CHOP, Toluca
- Netherlands (3):
  - Catharina Hospital, Eindhoven
  - Hagaziekenhuis, The Hague
  - Viecuri Medisch Centrum, Venlo
- North Macedonia (3):
  - PHI Clinical Hospital Dr Trifun Panovski Bitola, Bitola
  - Acibadem Sistina Hospital, Skopje
  - PHI University Clinic of Radiotherapy and Oncology, Skopje
- Peru (7):
  - Clinica San Antonio;Investigaciones Trujillo S.A.C., Trujillo, La Libertad
  - Hospital Nacional Daniel A Carrion, Bellavista
  - Hospital Militar Central, Jesus Maria
  - Hospital Central Fuerza Aerea Del Peru, Lima
  - Clínica Santa Beatriz, Lima
  - Oncologia S.A.C. - Instituto Peruano de Oncología & Radioterapia, Lima
  - Oncosalud Sac, Lima
- Philippines (9):
  - Saint Louis University Hospital of Sacred Heart, Baguio City, Benguet
  - University of Santo Tomas Hospital, Manila, National Capital Region
  - Riverside Medical Center, Inc., Bacolod City, Western Visayas (Region VI)
  - Baguio General Hospital and Medical Center, Baguio City
  - Metro Davao Medical and Research Center, Davao City
  - Cardinal Santos Medical Center, Manila
  - The Medical City, Pasig
  - East Avenue Medical Center, Quezon City
  - St. Luke's Medical Center - Quezon City, Quezon City
- Poland (8):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Szpital Morski Im. Pck, Gdynia
  - Narodowy Instytut Onkologii im. M.Sk?odowskiej-Curie - Pa?stwowy Instytut Badawczy Oddzia? Gliwice, Gliwice
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego, Grudziądz
  - Narodowy Instytut Onkologii - Panstwowy Instytut Badawczy, Oddzia? w Krakowie, Krakow
  - Centrum Terapii Wspolczesnej, Lodz
  - Centrum Onkologii Ziemi LUBELSKIEJ im. Sw Jana z Dukli, I oddz. Chemioterapii, Lublin
  - Centrum Medyczne Pratia, Poznan
- Portugal (10):
  - Unidade Local de Saude de Santa Maria, E.P.E. - Hospital de Santa Maria, Lisbon, Lisbon District
  - Hospital Senhora da Oliveira ? Guimaraes, E.P.E, Guimarães
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon
  - Champalimaud Cancer Center, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital Beatriz Angelo, Loures
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
  - Centro Hospitalar de Vila Nova de Gaia / Espinho E.P.E, Vila Nova de Gaia
  - Centro Hospitalar Trás Os Montes E Alto Douro EPE, Vila Real
- Romania (7):
  - Spitalul Clinic de Obstetrica si Ginecologie Filantropia, Bucure?ti
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Onco Clinic Consult SA, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Timisoara Emergency County Clinical Hospital, Timi?oara
- Serbia (5):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Health Center Kladovo, Kladovo
  - General Hospital Djordje Joanovic - Zrenjanin, Zrenjanin
- Slovakia (4):
  - Univerzitna nemocnica s poliklinikou Milosrdni bratia spol s r o, Bratislava
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, Košice
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (8):
  - Cape Town Oncology Trials, Cape Town
  - Cancercare Rondebosch Oncology, Cape Town
  - WITS Clinical Research Site PPDS, City of Johannesburg
  - Sandton Oncology Medical Group (Pty) Ltd, City of Johannesburg
  - Excellentis Clinical Trial Consultants, George
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Southern Cross Research South Africa (PTY) LTD, Mogale City
  - Wilgers Oncology Centre, Pretoria
- South Korea (17):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si, Chungcheongnam-do
  - Chungbuk National University Hospital, Cheongju-si
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - National Cancer Centre, Gyeonggi-do
  - CHA Bundang Medical Center, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Namdong-Gu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St. Mary?s Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Ulsan University Hosiptal, Songpa-Gu
  - Ajou University Hospital, Suwon
- Spain (61):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - ICO Badalona-H.U. Germans Trias i Pujol, Badalona, Barcelona
  - ALTHAIA Xarxa Assistencial de Manresa, Manresa, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital HM Nuestra Señora de la Esperanza, Santiago de Compostela, Burgos
  - Hospital de Jerez, Jerez de la Frontera, Cadiz
  - Consorcio Hospitalario Provincial de Castellon, Castellon de LA Plana/castello de LA Plana, Castellon
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario A Coruña, A Coruña, LA Coruna
  - CHUS H Clinico U de Santiago, Santiago de Compostela, LA Coruna
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitari Arnau de Vilanova, Lleida, Lerida
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - CHUVI ? H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Nuestra Senora de Valme, Seville, Sevilla
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario de Canarias, S. Cristobal de La Laguna, Tenerife
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario San Juan, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Clinica Tres Torres, Barcelona
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Reina Sofia, Córdoba
  - Institut Catala d'Oncologia Girona, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital General Universitario Gregorio Marañon, Madrid
  - IOB Madrid Institute of Oncology Hospital Beata Maria Ana de Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad Navarra, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - MD Anderson Cancer Center Madrid ? Espana, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario HM Sanchinarro ? CIOCC, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Sweden (5):
  - Länssjukhuset Ryhov, Jönköping
  - Södersjukhuset, Stockholm
  - Sundsvalls sjukhus, Sundsvall
  - Akademiska Sjukhuset, Uppsala
  - Västmanlands sjukhus Västerås, Västerås
- Switzerland (10):
  - Tumorzentrum Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Bern, Bern
  - Hirslanden Salem-Spital, Bern
  - Kantonsspital Graubünden KSGR, Chur
  - Luzerner Kantonsspital LUKS, Lucerne
  - Hirslanden Klinik St. Anna, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital STS AG Thun - Berner Oberland, Thun
  - Kantonsspital Winterthur Medizin Pneumologie, Winterthur
- Taiwan (11):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua County
  - Hsin-Chu Branch of National Taiwan University Hospital, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Cente, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
  - Taichung Veterans General Hospital, Xitun Dist.
- Thailand (3):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok Noi
- Turkey (Türkiye) (14):
  - Baskent Universitesi - Adana Uygulama Ve Arastirma Merkezi, Sariçam, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Fat?h
  - T.C. Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Izmir Medical Point Hospital, Izmir
  - Katip Celebi University- Izmir Ataturk Egitim ve Arastirma Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Arastirma ve Uygulama Hastanesi, Kocaeli
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Ac?badem Adana Hospital, Oncology Department, Seyhan/Adana
  - Acibadem Altunizade Hospital, Üsküdar
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Yen?mahalle
- Uganda (2):
  - Uganda Cancer Institute, Kampala
  - St Francis Hospital Nsambya, Kampala
- Ukraine (2):
  - Clinic Verum Expert LLC, Kyiv, KIEV Governorate
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
- United Kingdom (5):
  - Royal Sussex County Hospital, Brighton
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - Nottingham City Hospital, Nottingham
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing